CLINICAL TRIAL: NCT03312010
Title: A European, Prospective, Multi-Center, Double-Blind, Randomized, Controlled, Clinical Trial Investigating the Effects of High Frequency Peripheral Nerve Stimulation (PNS) in the Treatment of Chronic Back Pain
Brief Title: High Frequency PNS Stimulation Study for Back and Leg Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Curonix LLC (Industry)
Collaborators: AZ Delta (Other); GZA Ziekenhuizen Campus Sint-Augustinus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 30-004060
Record Dates: First submitted 2017-06-20; First posted 2017-10-17 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Chronic Back Pain; Chronic Back and Leg Pain

STUDY DESIGN:
Intervention Model Description: Prospective, partially double-blinded, randomized
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects and assessors randomized to HF blinded Subjects and assessors randomized to sham blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- High Frequency (Experimental): Subjects receiving high frequency pulse rate PNS treatment at T9 proximal peripheral nerves. Subjects and assessors blinded Randomization.
  Interventions: Device: PNS HF
- Sham (Sham Comparator): Subjects receiving Sham (non-active) PNS treatment at T9 proximal peripheral nerves. Subjects and assessors blinded to randomization. Subjects and assessors to be unblinded if pain scores are 30 mms or higher with VAS after 1-month follow-up. Upon this moment subjects to receive active stimulation
  Interventions: Device: PNS Sham

INTERVENTIONS:
Device: PNS HF — A needle and catheter is carefully inserted near your spinal column. The stimulator is then placed through the catheter and directed towards the T9 proximal peripheral nerves. The proximal end of the stimulator is then sutured underneath the skin of your back to the fascia to prevent migration.
  Arms: High Frequency
Device: PNS Sham — A needle and catheter is carefully inserted near your spinal column. The stimulator is then placed through the catheter and directed towards the T9 proximal peripheral nerves. The proximal end of the stimulator is then sutured underneath the skin of your back to the fascia to prevent migration.
  Arms: Sham

SUMMARY:
Prospective, double blinded, randomized, clinical study investigating the effects of high frequency PNS for the treatment of chronic back or back and leg pain.

DETAILED DESCRIPTION:
All subjects will have two permanent stimulators placed over the proximal peripheral nerves at T9 at the implant visit. The stimulators can easily be removed for non-responders. High frequency stimulation is typically programmed below sensory threshold. This type of stimulation lends itself to a placebo-controlled trial. For this study subjects will be randomized 1:1 at enrollment into a high frequency or sham group. Neither the subjects nor experimenters will be made aware of their randomization assignment for at least the first month of the trial. Subjects belonging to both groups will be unblinded to their assignment at the 1-month or a later visit (including unscheduled visit) if they have a VAS > 30 mms. Subjects belonging to the sham group will be reprogrammed with HF stimulation at this point. Subjects belonging to the HF stimulation group will keep stimulating with HF. Subjects reporting a VAS < 30 mms will continue to be blinded.

ELIGIBILITY:
Inclusion criteria

* Subject is ≥ 18 years of age at time of informed consent;
* Subjects have been diagnosed with predominant, chronic, intractable back pain with a VAS > 50 mm (on a 100-mm scale);
* Subjects have been diagnosed with predominant, chronic, intractable back pain for at least 6 months before study participation;
* Based on the medical opinion of the Principal Investigator, subject has a stable pain medication regiment;
* Based on the medical opinion of the Principal Investigator, there is no evidence of anatomic abnormalities that could jeopardize the placement of the device or pose a hazard to the subject;
* Subject is willing to undergo surgical implant procedure, attend visits as scheduled, and comply with the study requirements;
* Subject is willing and able to operate the patient programmer, recharging equipment and has the ability to undergo study assessments and provide accurate responses;
* Based on the opinion of the implanter, subject is a good surgical candidate for the implant procedure;
* Subject is male or non-pregnant female;
* Subject is deemed to be neuro-psycho-socially appropriate for implantation therapies based of the assessment of a clinical psychologist and principal investigator, using face-to-face encounters and the psychological testing described in the measures;
* Patient is capable of giving informed consent.

Exclusion criteria

* Obvious mechanical instability related to pain (diagnosed by imaging taken within the past 6 months);
* Unresolved malignancies in the last six months;
* Subject has post-herpetic neuralgia (shingles);
* Subject has an active systemic infection or is immune-compromised;
* Based on the medical opinion of the Principal Investigator the subject has other psychological conditions (e.g., psychosis, suicidal ideation, borderline personality disorder, somatization, narcissism), other health conditions (e.g., substance abuse, another chronic condition requiring the regular use of opioid medication), or other legal concerns that would preclude his/her enrollment in the study or potentially confound the results of the study;
* Subject is currently enrolled in or plans to enroll in any concurrent drug and/or device study while participating in this study;
* Insulin-dependent diabetic who is not controlled through diet and/or medication (determined by the physician) or non-insulin dependent diabetic who is not well controlled through diet and/or medication;
* Bleeding complications or coagulopathy issues;
* Pregnant/lactating or not using adequate birth control;
* A life expectancy of less than one year;
* Any active implanted device whether turned off or on;
* A previous PNS experience for the treatment of back pain;
* Conditions requiring Magnetic Resonance Imaging (MRI) evaluation or diathermy procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Responder rate | 1 month post-implant
  a > 50% reduction in back pain as measured by VAS with the Freedom PNS system in the HF (test) group as opposed to sham and conventional medical management

SECONDARY OUTCOMES:
VAS back pain | 1, 3, 6, 9, 12 and 36 months
  Percentage change from baseline in VAS for back pain
VAS leg pain | 1, 3, 6, 9, 12 and 36 months
  Percentage change from baseline in VAS for leg pain
ODI | 1, 3, 6, 9, 12 and 36 months
  Change from baseline in functionality using the ODI score

OTHER OUTCOMES:
PGIC | 1, 3, 6, 9, 12 and 36 months
  Subject satisfaction with the therapy as measured by the Patient Global Impression of Change (PGIC)
EQ-5D-5L | 1, 3, 6, 9, 12 and 36 months
  Changes from baseline in quality of life
AE's | 1, 3, 6, 9, 12 and 36 months
  Incidence of device related adverse events
Opioid Pain Medication | 1, 3, 6, 9, 12 and 36 months
  Prescribed opioid pain medications
Non-opioid Pain Medication | 1, 3, 6, 9, 12 and 36 months
  Prescribed non-opioid pain medication

CONTACTS AND LOCATIONS:
Locations (2):
- Belgium (2):
  - GZA Sint-Augustinus, Wilrijk, Antwerpen
  - AZ Delta, Roeselare

IPD SHARING:
Plan to Share IPD: No
Publication, Study outcomes

REFERENCES:
- [Derived] O'Connell NE, Ferraro MC, Gibson W, Rice AS, Vase L, Coyle D, Eccleston C. Implanted spinal neuromodulation interventions for chronic pain in adults. Cochrane Database Syst Rev. 2021 Dec 2;12(12):CD013756. doi: 10.1002/14651858.CD013756.pub2. PMID 34854473